CLINICAL TRIAL: NCT00045305
Title: A Phase II Study of Reduced Intensity Allogeneic Bone Marrow Transplant for the Treatment of Myelodysplastic Syndromes
Brief Title: Reduced-Intensity Regimen Before Donor Bone Marrow Transplant in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256928; E1902 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; refractory anemia; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Cyclosporine; Cyclosporins; Methotrexate; merphos; Photopheresis; Methoxsalen; Mycophenolic Acid; Pentostatin; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Preparative Regimen: Patients underwent photopheresis on two consecutive days and received pentostatin 4 mg/m2/d (total dose = 8 mg/m2) by continuous IV infusion on two consecutive days following photopheresis. Total body irradiation was administered on two consecutive days following pentostatin for a total of 600 cGy given in three 200 cGy fractionated doses.
  Transplantation: Unmanipulated allogeneic bone marrow or G-CSF mobilized peripheral blood stem cells were infused on day 0 within 48 hours of completion of TBI. Minimum cell dose was 2 ×106 CD34 cells/kg recipient.
  Acute graft-vs-host-disease (GVHD) prophylaxis: Patients received Cyclosporine or Tacrolimus per institutional preference or protocol beginning no later than day -1. Methotrexate (MTX) was administered on day +1 and +3. Mycofenolate mofetil (MMF) was introduced on day 100 and could be tapered and discontinued after 12 months if no active cGVHD.
  Interventions: Drug: Cyclosporine; Drug: Methotrexate; Drug: Photopheresis; Drug: Mycofenolate mofetil; Drug: Pentostatin; Procedure: allogeneic bone marrow; Procedure: peripheral blood stem cell; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Cyclosporine — Immunosuppressant
  Other Names: Sandimmune®; cyclosporin A; Neoral®Gengraf®; Gengraf®; CSA
Drug: Methotrexate — Antimetabolite
  Other Names: Methotrexate sodium; MTX; Mexate; Mexate-AQ; Folex; Folex PFS; Abitrexate; Rheumatrex; Amethopterin
Drug: Photopheresis — Psoralens
  Other Names: 8-methoxypsoralen; Uvadex ®; Methoxsalen
Drug: Mycofenolate mofetil — an antibiotic with immunosuppressamt properties isolated from Penicillium spp
  Other Names: Cellcept®; RS-61443; mycophenolic acid; Lilly-68618; MMF; Mycophenolate mofetil
Drug: Pentostatin — Purine analogue
  Other Names: DCF; 2-Deoxycoformycin; Nipent
Procedure: allogeneic bone marrow — Unmanipulated allogeneic bone marrow
Procedure: peripheral blood stem cell — G-CSF mobilized peripheral blood stem cell
Radiation: Total body irradiation — a total of 600 cGy given in 3 200 cGy fractionated doses
  Other Names: radiation therapy

SUMMARY:
RATIONALE: Photopheresis treats the patient's blood with drugs and ultraviolet light outside the body and kills the white blood cells. Giving photopheresis, pentostatin, and radiation therapy before a donor bone marrow or stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving pentostatin before transplant and cyclosporine or mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving pentostatin together with photopheresis and total-body irradiation work before donor bone marrow transplant in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate in patients with myelodysplastic syndromes treated with reduced-intensity allogeneic bone marrow transplantation, including photopheresis, total body irradiation, and pentostatin.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Determine the engraftment rate of donor cells in patients treated with this regimen.
* Determine the extent and duration of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a single-arm, two-stage, multicenter phase II study.

* Preparative Regimen: Patients undergo photopheresis using methoxsalen on days -7 and -6 and receive pentostatin intravenously (IV )continuously on days -5 and -4. Total body irradiation is administered on days -3 and -2 for a total of 3 doses.
* Transplantation: Allogeneic bone marrow or peripheral blood stem cells are infused on day 0.
* Acute graft-vs-host-disease (GVHD) prophylaxis: Patients receive cyclosporine IV on days -1 to 30 and then orally every 12 hours. Cyclosporine dose is then tapered beginning after day 50 and continuing for 6 months in the absence of GVHD. Once cyclosporine dose is significantly decreased, oral mycophenolate mofetil (MMF) is then administered twice a day. MMF dose is then tapered for 12 months in the absence of GVHD. Patients also receive methotrexate IV on days 1 and 3.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 33 patients would be accrued for this study within 2.1 years.

ELIGIBILITY:
Inclusion Criteria:

* One of the following cytologically proven myelodysplastic syndromes

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
  * RA with excess blasts
  * Chronic myelomonocytic leukemia
* International Prognosis Scoring System (IPSS) score of at least 0.5 OR red cell transfusion dependence for at least 6 months (2 units per month)

  * Patients with an IPSS score less than 0.5 may be eligible provided they previously had a higher IPSS score and received chemotherapy at that time
* Suitable human leukocyte antigen (HLA)-matched donor (related or unrelated) available

  * No cord blood donors
  * Related donors must be genotypically matched (HLA A, B and DR) at 5/6 or 6/6 loci and may be a sibling, parent, or child
  * Unrelated donors must have high resolution typing done at A, B, C and DR, and must be matched at all or may have a single antigen or allele mismatch at no more than one of these loci
* Patients must have < 20% blasts on bone marrow study within 1 month of study entry
* Age of 18 to 70 years
* Eastern Cooperative Oncology Group performance status 0-1
* Life expectancy at least 6 months
* At least 90 days since prior autologous bone marrow transplantation
* Serum erythropoietin level greater than 100 for patients who have not received a prior course of epoetin alfa
* No iron deficiency

  * Iron deficiency anemia treated with iron replacement therapy allowed
* Bilirubin less than 2.0 mg/dL
* Alkaline phosphatase less than 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3 times ULN
* Creatinine less than 2.0 mg/dL OR creatinine clearance greater than 50 mL/min
* Left ventricular ejection fraction (LVEF) at least 45% by Multigated Acquisition scan (MUGA) or echocardiogram
* Carbon Monoxide Diffusing Capacity (DLCO) at least 50% of predicted (corrected for hemoglobin)
* Forced expiratory volume in 1 second (FEV_1) at least 50% of predicted
* Recovered from prior chemotherapy
* Physically and psychologically capable of undergoing study regimen
* Able to receive 600 cGy of total body irradiation
* HIV negative
* Negative pregnancy test

Exclusion Criteria:

* Pregnant or nursing
* Having other medical condition that would reduce life expectancy
* Active ongoing infection
* Prior myeloablative or nonmyeloablative allogeneic transplantation for Myelodysplastic syndrome or acute myeloid leukemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10-24 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selina M. Luger, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (6):
- United States (6):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Jewish Hospital Cancer Center, Cincinnati, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was open to accrual on May 18, 2005 with the first patient accrued on October 24, 2006. By September 23, 2009, 17 patients were enrolled to the trial and the first 15 patients were included in the interim analysis. This trial did not meet pre-defined criteria to continue to the second stage. In the end, a total of 17 patients were enrolled to the trial from 7 participating institutions.
Period: Overall Study
Arm/Group | Arm I
Started | 17
Eligible and Treated | 17
Completed | 3
Not Completed | 14
Not completed — Lack of Efficacy | 6
Not completed — Adverse Event | 3
Not completed — Death | 3
Not completed — site error | 2

BASELINE CHARACTERISTICS:
Population: eligible and treated patients
Arm/Group | Arm I
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Completed response is defined as:
  Bone marrow evaluation: Repeat bone marrow showing < 5% myeloblasts with normal maturation of all cell lines, with no evidence for dysplasia (see dysplasia qualifier under peripheral blood evaluation).
  Peripheral blood evaluation [absolute values must last at least 2 months] Hemoglobin >11 g/dl (untransfused, not on erythropoietin) Neutrophils (1500/mm3 (not on a myeloid growth factor)) Platelets (100,000/mm3 (not on a thrombopoetic agent)) Blasts - 0% No dysplasia. No detectable cytogenetic abnormality, if preexisting abnormality was present
Time Frame: Monthly for the first 3 months from study entry, every 3 months for the first two years from study entry thereafter and then every 6 months for years 3-5.
Population: eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm I: Preparative Regimen: Patients underwent photopheresis on two consecutive days and received pentostatin 4 mg/m2/d (total dose = 8 mg/m2) by continuous IV infusion on two consecutive days following photopheresis. Total body irradiation was administered on two consecutive days following pentostatin for a total of 600 cGy given in three 200 cGy fractionated doses.
  Transplantation: Unmanipulated allogeneic bone marrow or G-CSF mobilized peripheral blood stem cells were infused on day 0 within 48 hours of completion of TBI. Minimum cell dose was 2 ×106 CD34 cells/kg recipient.
  Acute graft-vs-host-disease (GVHD) prophylaxis: Patients received Cyclosporine or Tacrolimus per institutional preference or protocol beginning no later than day -1. Methotrexate (MTX) was administered on day +1 and +3. Mycofenolate mofetil (MMF) was introduced on day 100 and could be tapered and discontinued after 12 months if no active cGVHD.
  Cyclosporine: Immunosuppressant
  Methotrexate: Antimetabolite
Arm/Group | Arm I
Number analyzed (Participants) | 17
percentage of participants | 35.3 [16.6 to 58.0]

2. Secondary Outcome: Number of Patients Who Developed Disease Progression After Achieving Complete Response
Description: Disease free survival (DFS) was listed as a secondary endpoint in the study protocol, which would be assessed in patients who achieved complete response (CR). It was defined to be time from CR to documented progression or to death without progression. Patients without documented progression or death reported were censored at the time of last disease evaluation. However, due to the small number of patients with CR, the number of patients who developed disease progression was reported here.
Time Frame: as for outcome 1
Population: eligible and treated patients who achieved complete response
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 6
participants | 1

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined to be the time from registration to death from any cause, with follow-up censored at the date of last contact. Kaplan-Meier method was used to estimate the distribution of OS.
Time Frame: as for outcome 1
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I
Number analyzed (Participants) | 17
years | 1.2 [0.5 to NA] — The upper bound of the 95% confidence interval has not reached yet for the median OS measure

4. Secondary Outcome: Proportion of Graft Versus Host Disease
Description: Proportion of Graft versus Host Disease is calculated as number of patients with Graft versus Host Disease divided by all eligible and treated patients
Time Frame: as for outcome 1
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I
Number analyzed (Participants) | 17
proportion of participants | 0.412 [0.184 to 0.671]

5. Secondary Outcome: Time to Engraftment for Neutrophil
Description: Time to neutrophil engraftment is defined from date of infusion to date of neutrophil engraftment. Neutrophil engraftment is defined as ANC > 500/mm3 on two consecutive measurements. The date of engraftment is the date of the first ANC > 500/mm3.
Time Frame: Daily while hospitalized and then at least 1x/week for the first 50 days and then at least every other week until day 100.
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I
Number analyzed (Participants) | 17
days | 18 [14 to 21]

6. Secondary Outcome: Time to Engraftment for Platelet
Description: Time to platelet engraftment is defined from date of infusion to date of platelet engraftment. The platelet engraftment is defined as platelets > 20,000 on two consecutive measurements, at least seven days apart, without platelet transfusions in between and for at least three days before the first measurement that is over 20,000. The date of engraftment is the date of the first measurement that is over 20,000.
Time Frame: as for outcome 5
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I
Number analyzed (Participants) | 17
days | 18 [16 to 30]

ADVERSE EVENTS:
Time Frame: Assessed at 30 days, 50 days, 100 days and 1 year post transplant
Description: Any severe (Grade ≥ 3) long term toxicity that the patient has experienced prior to diagnosis of progression/relapse that has not been previously reported would be collected via long-term follow up form at the following schedule: every 3 months for the first two years from study entry thereafter and then every 6 months for years 3-5
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 17/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
Anemia (Blood and lymphatic system disorders) | 14
Iron overload (Metabolism and nutrition disorders) | 1
White blood cell decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 17
Heart failure (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Fatigue (General disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 3
Enterocolitis infectious (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Infections and infestations - Other, spe (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - Other, spe (Infections and infestations) | 4
Edema limbs (General disorders) | 2
Alkaline phosphatase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 6
Creatinine increased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=17)
External ear inflammation (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 17
White blood cell decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 16
Electrocardiogram QT corrected interval (Investigations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 5
Insomnia (Psychiatric disorders) | 4
Chills (General disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Weight loss (Investigations) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Injection site reaction (General disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Cushingoid (Endocrine disorders) | 1
Hot flashes (Vascular disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Dysgeusia (Nervous system disorders) | 4
Vomiting (Gastrointestinal disorders) | 11
Hematuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations - Other, spe (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Edema limbs (General disorders) | 12
Edema trunk (General disorders) | 1
Alkaline phosphatase increased (Investigations) | 13
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 17
Creatinine increased (Investigations) | 16
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Sinus pain (Nervous system disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
General disorders and administration sit (General disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less